CLINICAL TRIAL: NCT00573469
Title: A Multicentre, Double-blind, Randomised, Parallel-group, Phase II Study to Assess Efficacy and Safety of D9421-C 9 mg and 15 mg Versus Placebo in Japanese Patients With Active Crohn's Disease
Brief Title: Efficacy and Safety Study of D9421-C 9 mg and 15 mg Versus Placebo in Japanese Patients With Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9421C00002
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Crohn's Disease
Keywords: gastrointestinal; GI; Crohn's disease; Japan; Japanese
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): D9421-C 9 mg
  Interventions: Drug: D9421-C, 9mg
- 2 (Active Comparator): D9421-C 15 mg
  Interventions: Drug: D9421-C, 15mg
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D9421-C, 9mg — D9421-C 9 mg was given once daily for 8 weeks.
  Arms: 1
Drug: D9421-C, 15mg — D9421-C 15 mg was given once daily for 8 weeks.
  Arms: 2
Drug: Placebo — D9421-C matching placebo was given once daily for 8 weeks.
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether treatment with D9421-C for 8 weeks in Japanese patients with mild to moderate active Crohn's disease will improve their symptoms of Crohn's disease and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged ≥ 18 and ≤ 65 years
* Diagnosis of Crohn's Disease

Exclusion Criteria:

* Having ileostomy or pouch and/or colostomy
* Having previous gastric surgery
* Having a known or suspected systemic infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Date, MD, PhD, Study Director — AstraZeneca
Locations (22):
- Japan (22):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Sakura, Chiba
  - Research Site, Chikushino-shi, Fukuoka
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kurume, Fukuoka
  - Research Site, Hashima-gun, Gifu
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kobe, Hyōgo
  - Research Site, Kyoto, Kyoto
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Osaka, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Tokorozawa, Saitama
  - Research Site, Shinjuku-ku, Tokyo
  - Research Site, Toyama, Toyama
  - Research Site, Itami
  - Research Site, Nishinomiya
  - Research Site, Tokyo

REFERENCES:
- [Derived] Suzuki Y, Motoya S, Takazoe M, Kosaka T, Date M, Nii M, Hibi T. Efficacy and tolerability of oral budesonide in Japanese patients with active Crohn's disease: a multicentre, double-blind, randomized, parallel-group Phase II study. J Crohns Colitis. 2013 Apr;7(3):239-47. doi: 10.1016/j.crohns.2012.06.006. Epub 2012 Jul 4. PMID 22766525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled on 16 October 2006. Last participant completed on 4 March 2008.
  Out of 90 screened participants, 77 participants (target was 75) were enrolled and included in Full Analysis set and safety analysis set. The numbers of participants in each set were 26 in D9421-C 9 mg, 25 in D9421-C 15 mg and 26 in Placebo, respectively.
Pre-assignment Details: Patients who had a CDAI score of less than 200 were excluded before randomisation.
Groups:
- D9421-C 9 mg: An enteric capsule including D9421-C 9 mg was given once daily.
- D9421-C 15 mg: An enteric capsule including D9421-C 15 mg was given once daily.
- Placebo: An enteric capsule without D9421-C was given once daily.
Period: Overall Study
Arm/Group | D9421-C 9 mg | D9421-C 15 mg | Placebo
Started | 26 | 25 | 26
Completed | 20 | 21 | 22
Not Completed | 6 | 4 | 4
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Other | 5 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D9421-C 9 mg | D9421-C 15 mg | Placebo | Total
Number analyzed (Participants) | 26 | 25 | 26 | 77
Age, Customized [Number; unit: Participants] — Age in Years
  Participants
    <30 years | 8 | 7 | 4 | 19.0
    >=30 years | 18 | 18 | 22 | 58.0
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 9 | 7 | 6 | 22.0
    Male | 17 | 18 | 20 | 55.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Remission of Crohn's Disease After 8-week Treatment
Description: Remission is defined by a Crohn's Disease Activity Index (CDAI) score of ≤ 150. That is, if a participant had 150 or less of CDAI score after 8-week treatment, the participant had the remission of Crohn's disease. The number of participants who had remission of Crohn's disease after 8-week treatment was the primary measure of this study.
Time Frame: Baseline to 8 weeks
Measure: Number; unit: Participants
Arm/Group | D9421-C 9 mg | D9421-C 15 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 26
Participants | 6 | 7 | 3

2. Secondary Outcome: Number of Participants Who Had Remission of Crohn's Disease After 2-week Treatment
Description: The number of participants who had remission of Crohn's disease (i.e., CDAI score ≤ 150) after 2-week treatment was one of the secondary measures of this study.
Time Frame: Baseline to 2 weeks
Measure: Number; unit: Participants
Arm/Group | D9421-C 9 mg | D9421-C 15 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 26
Participants | 2 | 3 | 0

3. Secondary Outcome: Number of Participants Who Had Remission of Crohn's Disease After 4-week Treatment
Description: as for outcome 2
Time Frame: Baseline to 4 weeks
Measure: Number; unit: Participants
Arm/Group | D9421-C 9 mg | D9421-C 15 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 26
Participants | 5 | 6 | 3

4. Secondary Outcome: Cumulative Percentage of Participants Who Achieved Remission up to 8 Weeks by Kaplan-Meier Method
Description: Time from randomisation to the remission of Crohn's disease defined as CDAI score  150 was analysed by Kaplan-Miere method. From this method, the cumulative percentage of participants who obtained up to 8 weeks were obtained.
Time Frame: At 8 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | D9421-C 9 mg | D9421-C 15 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 26
Percentage of participants | 38.5 (77.7) | 36.0 (84.7) | 19.0 (89.9)

5. Secondary Outcome: Change in CDAI Score From Baseline to 8 Weeks
Description: CDAI score is an index showing the condition of Crohn's disease and has no unit. The minimum is 0 and the maximum is not defined. Higher score shows worse condition and a decrease in score means improvement. In this study, participants who had 200 or higher of CDAI score were enrolled. The change from baseline to 8 weeks in CDAI score was measured.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | D9421-C 9 mg | D9421-C 15 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 26
Score on a scale | -48 (77.5) | -58 (84.7) | -27 (89.9)

ADVERSE EVENTS:
Arm/Group | D9421-C 9 mg | D9421-C 15 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/26 | 0/25 | 2/26
Other Adverse Events (participants affected / at risk) | 18/26 | 8/25 | 6/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D9421-C 9 mg (N=26) | D9421-C 15 mg (N=25) | Placebo (N=26)
Crohn's Disease (Gastrointestinal disorders) | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Perianal abscess (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | D9421-C 9 mg (N=26) | D9421-C 15 mg (N=25) | Placebo (N=26)
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Crohn's Disease (Gastrointestinal disorders) | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 0 | 2
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study without AZ approval before this study was completed.